CLINICAL TRIAL: NCT02957279
Title: A Cohort Study to Investigate the Impacts of Peripheral Blood Dendritic Cells-Derived Exosomes at Early Phase on the Prognosis in Human Sepsis
Brief Title: Dendritic Cells-Derived Exosomes in Human Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, President of department of surgery, Jinling Hospital, Jinling Hospital, China
Other Study IDs: 20161103
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Sepsis
Keywords: sepsis; exosomes; dendritic cell
MeSH Terms: conditions — Sepsis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral venous blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis group: The patients were admitted to the Jinling Hospital, who met the diagnosis of sepsis(Sepsis 3.0).
  Interventions: Drug: Antibiotics
- Healthy control group: Healthy volunteers.

INTERVENTIONS:
Drug: Antibiotics — In the sepsis group, antibiotics were used when needed.
  Groups: Sepsis group

SUMMARY:
The amount of peripheral blood exosomes has been confirmed to change in the endotoxin-induced infection. The primary objectives of this study are to compare the changes of peripheral blood dendritic cell-derived exosomes in the patients with sepsis and the healthy controls.

DETAILED DESCRIPTION:
This is a prospective, single-centered, clinical cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Patients were selected with the diagnostic standard "Sepsis 3.0".
* Healthy volunteers do not have serious illness.

Exclusion Criteria:

* Patients or volunteers do not agree to provide written informed consent and / or can not be legally authorized to provide informed consent.
* Patients give up treatments.
* Patients or volunteers withdrew from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were admitted to Jinling Hospital from November, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Amount of dendritic cell-derived exosomes | The first 4 hour after admission

SECONDARY OUTCOMES:
Compositions of microRNA in the dendritic cell-derived exosomes | The first 4 hour after admission

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Ren, MD, Principal Investigator — Jinling Hospital, Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China